CLINICAL TRIAL: NCT01054248
Title: A Randomised Open Label Trial Comparing Standard Dose of Dihydroartemisinin-piperaquine, Standard Fixed Artesunate-mefloquine Regimen and a Longer Regimen of Artemether-lumefantrine in the Treatment of Uncomplicated Malaria in Pregnancy
Brief Title: Randomised Trial of 3 Artemisinin Combination Therapy for Malaria in Pregnancy
Acronym: DMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMRU0905
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Malaria
Keywords: pregnancy, malaria, artemisinin, vivax, falciparum
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MAS3 (Experimental): Standard three day regimen of artesunate-mefloquine (12/24 mg/kg) given as artesunate 4mg/kg/day and mefloquine 8mg/kg/day on Days 0, 1 and 2.
  Interventions: Drug: Artesunate-mefloquine
- ALN+ (Active Comparator): Augmented 4 day regimen of artemether lumefantrine 2 doses per day for 4 days. Each dose consists of 5 tablets (20/120 mg of artemether/lumefantrine per tablet)
  Interventions: Drug: arthemeter-lumefantrin
- DP (Experimental): Standard 3 days regimen DHA-piperaquine: (DHA/PPQ 40 mg/320 mg) 2.4 mg/kg DHA and 20 mg/kg PPQ once daily for 3 days
  Interventions: Drug: dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine — Standard 3 days regimen DHA-piperaquine: (DHA/PPQ 40 mg/320 mg) 2.4 mg/kg DHA and 20 mg/kg PPQ once daily for 3 days
  Other Names: Artekin
  Arms: DP
Drug: Artesunate-mefloquine — Standard three day regimen of artesunate-mefloquine (12/24 mg/kg) given as artesunate 4mg/kg/day and mefloquine 8mg/kg/day on Days 0, 1 and 2.
  Arms: MAS3
Drug: arthemeter-lumefantrin — Augmented 4 day regimen of artemether lumefantrine 2 doses per day for 4 days. Each dose consists of 5 tablets (20/120 mg of artemether/lumefantrine per tablet).
  Other Names: Coartem
  Arms: ALN+

SUMMARY:
This is a randomised, open label trial, comparing standard dose of dihydroartemisinin-piperaquine (DP) with standard fixed artesunate-mefloquine regimen (MAS3) and with a longer regimen of artemether-lumefantrine (ALN+) in the treatment of uncomplicated malaria in pregnant women. The sample size is 335 women in each arm which would be 1005 women in total. Pregnant patients in 2nd and 3rd trimester with acute uncomplicated malaria who meet eligibility criteria will be asked to participate in the study. The primary objective is to determine if the efficacy of DP and MAS3 are superior to ALN+ in the treatment of uncomplicated malaria in pregnancy. The study will also incorporate a dense pharmacokinetic study of mefloquine and artesunate (15 women in the MAS3 arm) and a population pharmacokinetic study for mefloquine, piperaquine and lumefantrine.

DETAILED DESCRIPTION:
The 3 treatment regimens are 3 days of DHA-piperaquine (DP), 3 days of artesunate-mefloquine (MAS3) with mefloquine given as 8,8,8 mg/kg per day and an augmented dose of 4 days (5 tabs BID) of artemether- lumefantrine (ALN+). This will focus on efficacy and safety. Patients will be randomized equally to one of three treatment groups.

Within the trial there are two nested pharmacokinetic studies comprising dense data on 15 women for mefloquine and artesunate and sparse data for mefloquine, lumefantrine and piperaquine. Pregnant women will be followed up until delivery or day 63 if later than delivery and their infants will be followed until the end of the first year of life The follow up of babies will be monthly until 1 year (summarized in the table). Visits will include body weight, length, head circumference, arm circumference, physical examination, motor milestones by observation and caregiver interview, developmental examination and monthly haematocrit and stool testing. The mother is free to bring her infant at any time to the clinic and investigations appropriate to the presenting complaint and symptoms will be carried out as necessary to provide care for the infant.

Infants born to mothers who have a positive peripheral smear at delivery are at risk of congenital malaria and will be actively screened weekly for 2 months. In the last study one congenital malaria P.falciparum occurred at day 21 and the infant was very sick and was cured with artesunate. Infants who are positive for malaria would have a PCR spot to verify if the malaria was congenital.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Viable pregnancy of any gestation as assessed by ultrasound scanning
* Microscopically confirmed uncomplicated malaria (parasitaemia ≥ 5/500 WBC) with Plasmodium falciparum or Mixed infection (i.e. P.falciparum & P.vivax/ovale/malariae) or Plasmodium vivax/ovale/malariae
* Willingness and ability to comply with the study protocol for the duration of the trial
* Written informed consent provided
* No signs of labour

Additional criteria for patients in the detailed pharmacokinetic study group (N=24 in the MAS3 arm):

* HCT>25% (based on field reading i.e. capillary sample)
* P.falciparum monoinfection
* Agree to stay in the clinic for 7 days
* Written consent to participate the detailed PK subgroup

Exclusion Criteria:

* Known hypersensitivity to the study drugs
* P.falciparum asexual stage parasitaemia ≥ 4% RBCs
* Clinical or laboratory features of severe malaria based on WHO criteria-Appendix 1
* Gastrointestinal dysfunction that could alter absorption or motility
* History or known liver diseases or other chronic diseases (excluding thalassemia & G6PD deficiency)
* Presence of intercurrent illness or any condition which in the judgement of the investigator would place the patient at undue risk or interfere with the results of the study
* Splenectomy
* Hematocrit (HCT) <20% (based on field reading i.e. capillary sample) [ *NB: Dense mefloquine pharmacokinetic exclusion if HCT < 25%]
* Taking contraindicated medications
* History of narcotic or alcohol abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 511 (Actual)
Dates: Start 2010-02-16 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cure rate defined as clearance of asexual parasites without recurrence within the period between treatment and delivery or a 63 day period | Day 63 or until delivery, whichever occurs later

SECONDARY OUTCOMES:
Number of adverse events | Day 63
Biochemical and haematological changes | Day 28
Kinetic parameters of artesunate, mefloquine, piperaquine and lumefantrine | Day 42
Anaemia | Day 63
Gametocyte carriage | Day 63
Changes in the Reticulocyte counts | Day 63
Malaria infection rate at delivery and placental parasitaemia | Delivery
Pregnancy outcomes (abortions, low birth weight, premature birth, congenital abnormality, stillbirths, neonatal and infant mortality) | Delivery
Infant growth and development at 1 year of life | 1 year after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rose McGready, MBBS, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Derived] Saito M, Wilaisrisak P, Pimanpanarak M, Viladpai-Nguen J, Paw MK, Koesukwiwat U, Tarning J, White NJ, Nosten F, McGready R. Comparison of lumefantrine, mefloquine, and piperaquine concentrations between capillary plasma and venous plasma samples in pregnant women with uncomplicated falciparum and vivax malaria. Antimicrob Agents Chemother. 2024 May 2;68(5):e0009324. doi: 10.1128/aac.00093-24. Epub 2024 Apr 10. PMID 38597636
- [Derived] Saito M, Carrara VI, Gilder ME, Min AM, Tun NW, Pimanpanarak M, Viladpai-Nguen J, Paw MK, Haohankhunnatham W, Konghahong K, Phyo AP, Chu C, Turner C, Lee SJ, Duanguppama J, Imwong M, Bancone G, Proux S, Singhasivanon P, White NJ, Nosten F, McGready R. A randomized controlled trial of dihydroartemisinin-piperaquine, artesunate-mefloquine and extended artemether-lumefantrine treatments for malaria in pregnancy on the Thailand-Myanmar border. BMC Med. 2021 Jun 10;19(1):132. doi: 10.1186/s12916-021-02002-8. PMID 34107963